CLINICAL TRIAL: NCT02393729
Title: Functional MRI Study of the Involvement of Cortico-cerebellar and Cortico-striatal Networks in Children With a Developmental Coordination Disorder (DCD) and/or Developmental Dyslexia (DD)
Brief Title: Functional MRI Study in Children With a Developmental Coordination Disorder (DCD) and/or Developmental Dyslexia (DD)
Acronym: FMRI-DCD-DD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 10 155 02; N°RCB : 2010-A00909-30 (Registry Identifier: ANSM)
Record Dates: First submitted 2015-03-13; First posted 2015-03-19 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Developmental Dyslexia; Developmental Coordination Disorder
MeSH Terms: conditions — Dyslexia; Motor Skills Disorders | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- children with DCD (Other): Children with Developmental Coordination Disorder (DCD) will have neuropsychological assessment and MRI study
  Interventions: Behavioral: Neuropsychological assessment; Other: MRI Study
- children with DD (Other): Children with Developmental Dyslexia (DD) will have neuropsychological assessment and MRI study
  Interventions: Behavioral: Neuropsychological assessment; Other: MRI Study
- children with DCD + DD (Other): Neuropsychological assessment and MRI study
  Interventions: Behavioral: Neuropsychological assessment; Other: MRI Study
- control children (Other): Neuropsychological assessment and MRI study
  Interventions: Behavioral: Neuropsychological assessment; Other: MRI Study

INTERVENTIONS:
Behavioral: Neuropsychological assessment — The neuropsychological assessment will include an assessment of:
  * Intellectual ability
  * Laterality
  * Reading Skills
  * Motor skills
  * Oral Language
  * Attention
  * Child's behaviour
Other: MRI Study — It will include a first session of about an hour outside MRI for familiarization with the environment of the MRI. The MRI will then be made after a break of 15 minutes
  * Morphological time: this time include the initial acquisition of a sequence of anatomical 3D T1-weighted high-resolution contiguous axial slices and the imaging of diffusion tensor.
  * Functional time: The experimental paradigm is a paradigm as a block with alternating phase of motor and rest conditions. The two motor tasks are: a Learning motor sequence or motor sequence task and Automated motor sequence or AT (automated task).
  Other Names: structural and functional MRI

SUMMARY:
All the studies underlined the high frequency of co-morbid associations in specific learning disorders. Understanding the reasons for these associations could enable us to determine the cerebral bases that underlie each disorder. Their frequent association suggests the etiological bases are partly common, it seems logical to turn to explanatory models of various common specific disorders. The model recently proposed by Nicholson & Fawcett (2007) suggests a specific disorder of procedural learning. But the brain networks involved in this learning could be achieved separately. We intend therefore to study the neural networks involved in learning procedural and compare networks recruited among children with specific learning disorder alone or in combination (co-morbidity). The children included in the study have either a Developmental Dyslexia or a Developmental Coordination Disorder, or both. The procedure includes a neuropsychological evaluation and a brain MRI study with a morphological and a functional part. During fMRI the child realizes a automated motor task contrasting with a task involving learning procedural.

ELIGIBILITY:
Inclusion criteria:

These children presenting either a specific disorder in learning to read (developmental dyslexia or DD) type phonological or mixed as defined by World Health Organisation or a Developmental Coordination Disorder (DCD) as defined by Diagnostic and Statistical Manual IV criteria or the association of both disorders (DCD + DD).

Or in the control group:

Children having no neurological or psychiatric disorder, mental retardation with IQ (Intelligence quotient) > 70 and DCD (score> 15 percentile on the Movement ABC) and Dyslexia (reading delay should not exceed 12 months) The age of children included in the study is between 8 and 12 years. The inclusion of subjects from 8 years is justified to have an optimal level of cooperation of the child in the MRI, in order to determine the status of children for reading and the fact that most of validated neuropsychological tests for reading are for the age 8 to 12 years.

Children and their parents must have given their free and informed consent signed. The representative of the child shall be affiliated to a social security scheme.

The children included in the study will be all right handed.

Exclusion criteria:

Mental retardation as defined by DSM IV criteria by an estimated IQ from the Wechsler scales less than 70.

The presence of a Specific Language Impairment (or dysphasia): a score below -2 SD (standard deviation) in at least one of three tests for language assessment is a criterion for exclusion.

The presence of a dyslexia-type surface defined by a specific disorder in learning to read without difficulty for metaphonological tests and/or an exclusive impairment of the addressing reading route (reading irregular words).

Children regularly practicing a musical instrument conferring a high manual dexterity such as piano or guitar.

Children with neurological or psychiatric disorders as epilepsy for example. Children under psychotropic medication such as anticonvulsant. Treatment with methylphenidate is not an exclusion criterion but treatment should be discontinued at least 48 hours before performing MRI. Children with ADHD according to DSM IV criteria.

The presence of a cons-indication for a MRI.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2011-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
difference in the level of brain activity | 1 day
  The difference in the level of brain activity obtained by contrasting the result of the automated task and that task with learning in the same patient-adjusted performance.
The level of brain activity obtained by fMRI | 1 day
  The level of brain activity obtained by fMRI will be estimated by the blood flow in milliliters per minute using a standardized procedure and validated specific MRI used and managed entirely by dedicated software (SPM8 - Welcome Department of Cognitive Neurology, London, UK). The performance adjustment is made in the analysis of the estimated difference in blood flow using a mixed model. Regions of interest are the primary motor cortex, the supplementary motor area, the pre motor cortex, the striatum and the cerebellum. These regions will be studied in both hemispheres.

SECONDARY OUTCOMES:
The performance of subjects | 1 day
  The performance of subjects evaluated in terms of frequency of movements in Hz and the number of erroneous restraints. The average frequency of movements for each block will be used as a covariate in the statistical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Yves Chaix, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Hôpital des Enfants, Toulouse, France

REFERENCES:
- [Result] Biotteau M, Peran P, Vayssiere N, Tallet J, Albaret JM, Chaix Y. Neural changes associated to procedural learning and automatization process in Developmental Coordination Disorder and/or Developmental Dyslexia. Eur J Paediatr Neurol. 2017 Mar;21(2):286-299. doi: 10.1016/j.ejpn.2016.07.025. Epub 2016 Aug 12. PMID 27546352
- [Result] Biotteau M, Albaret JM, Lelong S, Chaix Y. Neuropsychological status of French children with developmental dyslexia and/or developmental coordination disorder: Are both necessarily worse than one? Child Neuropsychol. 2017 May;23(4):422-441. doi: 10.1080/09297049.2015.1127339. Epub 2016 Jan 4. PMID 26729293